CLINICAL TRIAL: NCT03013426
Title: A Phase Ib, Dose-finding and Pharmacodynamic Study of NVX-508 in Sickle Cell Disease Patients
Brief Title: A Phase Ib Study of NVX-508 in Sickle Cell Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: NuvOx Pharma suspended the clinical program related to this study.
Sponsor: Amma Owusu-Ansah, MD (Other)
Collaborators: NuvOx LLC (Industry); Noguchi Memorial Institute for Medical Research (Other)
Responsible Party: Sponsor-Investigator, Amma Owusu-Ansah, MD, Assistant Professor of Medicine and Clinical Director, Center for Translational and International Hematology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO16110118
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NVX-508 (Experimental): Administration of 1, 2 or 4 doses of NVX-508 at three dose levels; 0.05ml/kg. 0.1ml/kg and 0.17ml/kg in a 3 + 3 design.
  Interventions: Drug: NVX-508

INTERVENTIONS:
Drug: NVX-508 — Administration of NVX-508 emulsion intravenously

SUMMARY:
This Phase 1b study in adults with sickle cell disease (SCD) in steady-state (non-acutely ill) aims to evaluate safety and toxicity of NVX-508 in a multi-dosing paradigm as well as to determine the maximum tolerated dose (MTD) in this population. The information gained from this study will be used in making decisions about the appropriate dose(s) and dosing schedule in future multicenter studies of the efficacy of NVX-508 in the treatment of vaso-occlusive episodes (VOE).

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a genetic disorder of hemoglobin that affects millions of individuals worldwide, with sub-Saharan Africa bearing the greatest burden of disease. The leading causes of hospitalization and death in individuals with sickle cell disease are painful VOE (associated with tissue injury from reduced oxygen supply) and "acute chest syndrome" respectively. Acute chest syndrome (ACS) is a form of acute lung injury unique to SCD that arises de novo or during the course of painful VOE.

A safe, reliable therapeutic deployed early in the course of painful VOE (with or without ACS) that restores oxygen supply to tissues, could potentially attenuate tissue injury, resolve pain and improve patient outcomes.

NVX-508 is a liquid fluorocarbon which transports oxygen. Stoichiometrically, NVX-508 has 200 times the oxygen carrying capacity of human hemoglobin.Oxygen is taken up by NVX-508 as it circulates through the alveolar capillary bed in the lungs and is released in blood and tissues with low oxygen content. Consequently, if it were administered intravenously (IV) and passed through the lungs of patients, it would take up oxygen, increasing the oxygen concentration in blood in a dose-dependent manner and release it to tissues with low oxygen.

The active component of NVX-508 was originally developed as an ultrasound contrast agent. It has been tested as such in over 2200 patients to whom it was safely administered as a bolus IV injection.The pharmacokinetics of NVX-508 in humans exhibits a biphasic decline after an iv bolus dose; a rapid initial decline followed by a slow terminal phase. The terminal phase t1/2 (half- life) ranges from 81-99.5 min for doses of 0.15-0.35 ml/kg. NVX-508 is not metabolized in humans, it is removed from the body unchanged in the breath (expired air) .

The rationale for studying NVX-508 for SCD is based on data from preclinical studies in the mouse model of ACS. NVX-508 when used as rescue therapy in the mouse model, restored oxygen saturation to baseline in mice experiencing hypoxemia, with 100% survival. NVX-508 reduced pulmonary vascular congestion in SCD mice experiencing ACS.

Hypothesis: Intravenous delivery of 4 doses of NVX-508 of up to 0.17 ml/kg per dose, infused over 30 minutes will be well tolerated.

Experimental design: Dose-ranging study in adults with diagnosis of SCD (SS, SC, S-Beta + thalassemia, S-Beta0 thalassemia, and SS/S-Hemoglobin D (SD)or S in combination with another variant hemoglobin) , who are in steady state (no painful episode, hospitalization or blood transfusion in the preceding 4 weeks) will be recruited from a single institution (Ghana Institute of Clinical Genetics, Korle-Bu, Accra, Ghana) to participate in the study.

The study has a 3 + 3 design. The first cohort of 3 subjects enrolled in the study shall be administered one dose (0.05 mL/kg) of NVX-508, the next cohort of 3 will be treated using two doses of NVX-508 at 0.05 mL/kg and subsequent cohort will be assigned to four doses of NVX-508. Higher doses of 0.1ml/kg and 0.17ml/kg will be administered Intra-patient dose escalation will not be allowed. Each dose shall be administered as slow IV push over 5-10 minutes with the next dose administered no less than 90 minutes after cessation of the prior infusion, but not more than 120 minutes later.

Within each cohort, when the first subject is treated, there will be a 72 hour observation interval before the next two subjects are treated at the same dose.

Study Procedures

A maximum of 24 adults with sickle cell disease aged 18 years and above will be recruited into the study.

Screening - After giving informed consent, potential study participants will undergo screening which comprises a standardized history and physical examination, lab tests (blood counts, serum chemistries) and electrocardiogram( EKG). Eligible participants will return within a week to be enrolled in the study.

Intervention - Study participants will go to a designated staffed phase I center for administration of the study drug. They will have baseline evaluations (arterial blood gas evaluation, hemoglobin and EKG) done prior to administration of the study drug. They will receive 1, 2 or 4 doses of the study drug depending They will be continuously monitored by medical research staff and the principal investigator prior to, during and in the 4 hour observation period post intervention, with physical examination, labs ( complete blood counts, serum chemistries, coagulation profile and blood samples drawn for blood gas evaluation and EKGs.

Subjects will be discharged from the clinical trials facility after the 4 hour observation period if they have had no adverse events requiring further clinical management. There will be a one week post-intervention observation period for dose-limiting toxicity for each subject, at the end of which they will have a follow up visit.

Follow up - 1 week after administration of NVX-508, subjects will have a follow-up visit at the clinical trial facility which includes history, physical exam and labs. If there are no adverse events or problems requiring continued clinical care and monitoring, subjects will exit the study once the lab and clinical data from the visit have been completely reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SCD without acute VOE and/or ACS.
* Age 18 years and older
* Adequate hematologic, renal and hepatic function, defined by:

  1. Absolute neutrophil count (ANC) ≥ 1.5 x109/L
  2. Platelet count ≥ 100 x 109/L,
  3. Hemoglobin ≥ 60 g/L
  4. International normalized ratio (INR) < 1.5 x upper limit of normal (ULN)
  5. Activated partial thromboplastin time (APTT) < 1.5 x ULN
  6. Plasma creatinine < 1.5 x ULN
  7. Total bilirubin < 2.5 x ULN (in the presence of Gilbert's syndrome or indirect hyperbilirubinemia caused by hemolysis)
  8. Aspartate transaminase (AST) < 2.5 x ULN
  9. Alanine transaminase (ALT) < 2.5 x ULN
* Ability of the prospective subject to understand and willingness to sign written informed consent document

Exclusion Criteria:

* Patients who have received any other investigational agent within 4 weeks before enrollment.
* Patients who have had a VOE/ACS in the previous 4 weeks before enrollment.
* Stroke or transient ischemic attack within 6 months before enrollment.
* Myocardial infarction within 6 months before enrollment, unstable angina, New York Heart Association class II or greater congestive heart failure, or uncontrolled hypertension (systolic BP > 160 mmHg and/or diastolic BP > 100 mmHg).
* Congenital long QT syndrome, or corrected QT interval ( QTc) > 450 milliseconds (msec) in males and > 470 mSec in females on EKG.
* Uncontrolled arrhythmia or any history of clinically significant arrhythmia in the past 6 months
* Clinically-significant chronic obstructive pulmonary disease or asthma that is not controlled by medication.
* A history of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer or other solid tumors curatively treated with no evidence of disease for ≥ 2 years.
* Current anticoagulant or antiplatelet therapy, except for prophylactic doses of low molecular weight heparins or low-dose aspirin.
* History of allergic reactions attributed to compounds of similar chemical composition to NVX- 508.
* Women who are pregnant or breastfeeding.
* Inability to comply with study procedures.
* History or evidence of any other clinically-significant condition that, in the opinion of the investigator, would pose a risk to subject safety or interfere with study procedures, evaluation or completion.
* Patients with active VOE or ACS or other significant current acute complication of SCD.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of NVX-508 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amma T Owusu-Ansah, MD, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modell B, Darlison M. Global epidemiology of haemoglobin disorders and derived service indicators. Bull World Health Organ. 2008 Jun;86(6):480-7. doi: 10.2471/blt.06.036673. PMID 18568278
- [Background] Grosse SD, Odame I, Atrash HK, Amendah DD, Piel FB, Williams TN. Sickle cell disease in Africa: a neglected cause of early childhood mortality. Am J Prev Med. 2011 Dec;41(6 Suppl 4):S398-405. doi: 10.1016/j.amepre.2011.09.013. PMID 22099364
- [Background] Johnson JL, Dolezal MC, Kerschen A, Matsunaga TO, Unger EC. In vitro comparison of dodecafluoropentane (DDFP), perfluorodecalin (PFD), and perfluoroctylbromide (PFOB) in the facilitation of oxygen exchange. Artif Cells Blood Substit Immobil Biotechnol. 2009;37(4):156-62. doi: 10.1080/10731190903043192. Epub 2009 Jun 22. PMID 19548131
- [Background] Riess JG. Understanding the fundamentals of perfluorocarbons and perfluorocarbon emulsions relevant to in vivo oxygen delivery. Artif Cells Blood Substit Immobil Biotechnol. 2005;33(1):47-63. doi: 10.1081/bio-200046659. PMID 15768565
- [Background] Grayburn PA, Weiss JL, Hack TC, Klodas E, Raichlen JS, Vannan MA, Klein AL, Kitzman DW, Chrysant SG, Cohen JL, Abrahamson D, Foster E, Perez JE, Aurigemma GP, Panza JA, Picard MH, Byrd BF 3rd, Segar DS, Jacobson SA, Sahn DJ, DeMaria AN. Phase III multicenter trial comparing the efficacy of 2% dodecafluoropentane emulsion (EchoGen) and sonicated 5% human albumin (Albunex) as ultrasound contrast agents in patients with suboptimal echocardiograms. J Am Coll Cardiol. 1998 Jul;32(1):230-6. doi: 10.1016/s0735-1097(98)00219-8. PMID 9669275
- [Background] Correas JM, Meuter AR, Singlas E, Kessler DR, Worah D, Quay SC. Human pharmacokinetics of a perfluorocarbon ultrasound contrast agent evaluated with gas chromatography. Ultrasound Med Biol. 2001 Apr;27(4):565-70. doi: 10.1016/s0301-5629(00)00363-x. PMID 11368867